CLINICAL TRIAL: NCT02663232
Title: Epidemiological Study of V600 BRAF Mutation in Spanish Patients Diagnosed With Metastatic Melanoma: ABSOLUT-BRAF Study
Brief Title: Study to Analyze Mutations in V600 BRAF Oncogen in Participants With Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30089
Record Dates: First submitted 2015-11-20; First posted 2016-01-26 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Cancers
Keywords: V600 BRAF mutation; Metastatic melanoma
MeSH Terms: conditions — Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Metastatic melanoma: Participants with metastatic melanoma who attend their physicians during the 18-month recruitment period and have valid biological samples available for BRAF mutation testing will be included in the study. There will be no intervention in this study.

SUMMARY:
This is a national, multicenter, cross-sectional epidemiological study in adult Spanish participants diagnosed with advanced or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Valid tumor samples from participants diagnosed with Stage IIIc or IV melanoma
* Written informed consent granted

Exclusion Criteria:

- Do not fulfill one or more inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with metastatic melanoma who have valid samples for BRAF mutation testing and give their informed consent will be included in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- Spain (25):
  - Palma de Mallorca, Balearic Islands
  - Jerez de la Frontera, Cadiz
  - Santander, Cantabria
  - Castellon, Castellon
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña, LA Coruña
  - Cartagena (Murcia), Murcia
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Santa Cruz de Tenerife, Tenerife
  - Bilbao, Vizcaya
  - Barcelona
  - Burgos
  - Cáceres
  - Girona
  - Granada
  - Lleida
  - Madrid
  - Málaga
  - Murcia
  - Salamanca
  - Seville
  - Toledo
  - Valencia
  - Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Metastatic Melanoma: Participants with metastatic melanoma who attended their physicians during the 18-month recruitment period and had valid biological samples available for BRAF mutation testing were included in the study. There was no intervention in this study.
Period: Overall Study
Arm/Group | Metastatic Melanoma
Started | 264
Completed | 264
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study were included in the analysis.
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
Age, Continuous [Median (Full Range); unit: years] | 68.0 [56.0 to 77.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With V600 BRAF Mutation Status
Description: Presence or absence of mutations in the V600 BRAF oncogene was determined in all eligible participants. Data collection and management of BRAF mutation testing was carried out using the Biomarker point® online platform. The platform was used as an electronic case report form (e-CRF) for collecting information in electronic format via a website. Percentage of participants with BRAF mutation status (mutated BRAF, wild type, not available) were reported.
Time Frame: Day 1
Population: All enrolled participants were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Mutated BRAF | 41.3 [35.3 to 47.5]
  Wild type | 58.3 [52.1 to 64.3]
  Not available | 0.4 [0.02 to 2.4]

2. Secondary Outcome: Percentage of Participants Categorized by Melanoma Stage
Description: Melanoma stages were categorized (according to American Joint Committee on Cancer [AJCC]) as IIIc (advanced stage of melanoma), M1a (metastases to skin, subcutaneous, or distant lymph nodes, normal lactate dehydrogenase (LDH) level, M1b (lung metastases, normal LDH) and M1c (metastases to all other visceral sites and normal LDH or distant metastases to any site combined with an elevated serum LDH level). Of these Stage IIIc was used as the referral category for comparisons.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  IIIc | 14.4
  M1a | 19.3
  M1b | 13.3
  M1c | 22.7
  Missing data | 29.9
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of Melanoma Stage (IIIC [referral category] versus (vs) M1a vs M1b vs M1c) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.001, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation
Statistical Analysis 2: Comparison: Metastatic Melanoma; The association of Melanoma Stage IIIC/M1a/M1b [referral category] vs M1c with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.196, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation
Statistical Analysis 3: Comparison: Metastatic Melanoma; The association of Melanoma Stage IIIc with the risk of BRAF mutation (Yes/No) was assessed using multivariate regression analysis; Test type: Superiority or Other; p = 0.002, Multivariate regression analysis; Multivariate regression analysis of clinical risk factors for BRAF mutation
Statistical Analysis 4: Comparison: Metastatic Melanoma; The association of Melanoma Stage M1a (using Melanoma Stage IIIC as referral category) with the risk of BRAF mutation (Yes/No) was assessed using multivariate regression analysis; Test type: Superiority or Other; p = 0.028, Multivariate regression analysis; Multivariate regression analysis of clinical risk factors for BRAF mutation (n=184); Hazard Ratio (HR) = 2.716, 95% CI 2-sided [1.115 to 6.616]
Statistical Analysis 5: Comparison: Metastatic Melanoma; The association of Melanoma Stage M1b (using Melanoma Stage IIIC as referral category) with the risk of BRAF mutation (Yes/No) was assessed using multivariate regression analysis; Test type: Superiority or Other; p = 0.142, Multivariate regression analysis; Multivariate regression analysis of clinical risk factors for BRAF mutation (n=184); Hazard Ratio (HR) = 0.466, 95% CI 2-sided [0.168 to 1.291]
Statistical Analysis 6: Comparison: Metastatic Melanoma; The association of Melanoma Stage M1c (using Melanoma Stage IIIC as referral category) with the risk of BRAF mutation (Yes/No) was assessed using multivariate regression analysis; Test type: Superiority or Other; p = 0.653, Multivariate regression analysis; Multivariate regression analysis of clinical risk factors for BRAF mutation (n=184); Hazard Ratio (HR) = 0.822, 95% CI 2-sided [0.351 to 1.928]

3. Secondary Outcome: Percentage of Participants With Family History of Melanoma
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants | 5.7
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of Family family history of melanoma (yes vs no) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.240, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation

4. Secondary Outcome: Percentage of Participants With Sun Exposure
Description: Data were obtained to classify the population with sun exposure as those with low, intermittent or chronic exposure. For the sub-analysis of low, intermittent and chronic exposure, percentages were calculated based on the population with any sun exposure.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Any exposure (n=264) | 49.2
  Low exposure (n=130) | 12.3
  Intermittent exposure (n=130) | 60.8
  Chronic exposure (n=130) | 26.9
  Missing data (n=264) | 13.6
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of sun exposure yes vs no with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.719, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation

5. Secondary Outcome: Percentage of Participants Categorized by Primary Tumor Location
Description: Primary tumor location included limbs (upper and lower extremities), trunk, head/neck, mucosa, uveal, acral, other (other than these specified locations), unknown (exact location unknown), and not available.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Limbs (Upper extremities) | 9.1
  Limbs (Lower extremities) | 22.0
  Trunk | 28.4
  Head/Neck | 14.4
  Mucosa | 6.8
  Uveal | 4.2
  Acral | 1.1
  Other | 0.4
  Unknown | 8.7
  Not available | 6.1
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of primary tumor site (trunk [referral category] vs head and neck vs upper extremities vs lower extremities vs. visceral/mucosa) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.262, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation

6. Secondary Outcome: Percentage of Participants Categorized By LDH Level
Description: Normal LDH levels range from 140 units per liter (U/L) to 280 U/L.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Normal | 20.1
  High | 51.5
  Unknown | 28.4
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of LDH (elevated [referral category] vs normal vs unknown) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.313, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation

7. Secondary Outcome: Median Time Since Diagnosis of Melanoma
Description: Median time from the diagnosis of primary melanoma to advanced disease was determined in years.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis except for one participant with missing data.
Measure: Median (Full Range); unit: years
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 263
years | 1.0 [0.1 to 3.3]
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of time since diagnosis of primary melanoma (continuous variable) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.291, Bivariate regression analysis; Bivariate regression analysis of clinical risk factors for BRAF mutation

8. Secondary Outcome: Percentage of Participants Categorized by Tumor Sample Source (Primary Tumor or Metastatic Sites)
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Metastases | 62.9
  Primary tumor | 34.1
  Relapses | 2.3
  Unknown | 0.8
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of tumor sample source (primary tumor [referral category] vs metastases vs relapses) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.164, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

9. Secondary Outcome: Percentage of Participants Categorized by Tumor Sample Type (Paraffin-embedded Tissue Blocks, Paraffin Block Slides, Cytology Slides, or Other)
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Paraffin-embedded blocks | 73.5
  Slides of paraffin blocks | 22.3
  Cytological slides | 3.4
  Other | 0.8
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of tumor sample type (paraffin-embedded blocks [referral category] vs slides of paraffin blocks vs cytology slides) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.505, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

10. Secondary Outcome: Percentage of Participants Categorized by Method of Fixation (Buffered Formalin or Others)
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Buffered formalin | 92.8
  Other | 5.3
  Unknown | 1.9
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of method of fixation (buffered formalin [referral category] vs other) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.701, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

11. Secondary Outcome: Percentage of Participants Categorized by Breslow Thickness
Description: Breslow thickness is defined as the total vertical height of the melanoma, from the very top (called the granular layer) to the area of deepest penetration in the skin. An instrument called an ocular micrometer is used to measure the thickness of the excised (removed) tumor. In general, the higher the Breslow thickness, the worse the prognosis. The classifications were lesser than or equal to (≤) 1.0 millimeters (mm), 1.01 - 2.0 mm, 2.01 - 4.0 mm, greater than (>) 4.0 mm and Unknown.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  ≤1 mm | 5.7
  1.01 - 2.0 mm | 14.4
  2.01 - 4.0 mm | 22.3
  >4 mm | 27.3
  Unknown | 30.3
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of Berslow thickness (≤1 mm [referral category] vs 1.01-2 mm vs 2.01-4 mm vs 4 mm) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.683, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

12. Secondary Outcome: Percentage of Participants With Ulceration
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  With ulceration | 41.7
  Without ulceration | 26.1
  Unknown | 32.2
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of Ulceration (no [referral category] vs yes) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.615, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

13. Secondary Outcome: Percentage of Participants With Regression
Description: Regression in melanoma is the replacement of tumor tissue with fibrosis, degenerated melanoma cells, lymphocytic proliferation, and telangiectasia formation.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  With regression | 9.5
  Without regression | 53.0
  Unknown | 37.5
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of presence of regression (Without regression [referral category] vs With regression) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.949, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

14. Secondary Outcome: Percentage of Participants With Vascular Invasion
Description: Vascular invasion is defined as the appearance of cancer cells in the lymphatic and blood streams.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  With vascular invasion | 8.3
  Without vascular invasion | 58.7
  Unknown | 33.0
Statistical Analysis 1: Comparison: Metastatic Melanoma; The association of Vascular invasion (Without vascular invasion [referral category] vs With vascular invasion) with the risk of BRAF mutation (Yes/No) was assessed using bivariate regression analysis; Test type: Superiority or Other; p = 0.374, Bivariate regression analysis; Bivariate regression analysis of anatomopathological risk factors for BRAF mutation

15. Secondary Outcome: Percentage of Participants Categorized by Method of DNA Extraction (Cobas® BRAF V600 Mutation Test or Others)
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Cobas® BRAF V600 Mutation Test | 93.1
  Other | 6.8

16. Secondary Outcome: Percentage of Participants Categorized by Method of BRAF Mutation Testing (Cobas® 4800 BRAF V600 Mutation Test or Others)
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  Cobas® 4800 BRAF V600 Mutation Test | 96.2
  Other | 3.8

17. Secondary Outcome: Percentage Participants Categorized by the Percentage of Tumor Cells Referred to the Technique
Description: The samples were classified based on the percentage of tumor cells referred to the technique as follows: <60 percent (%), 60-80%, >80% and Unknown.
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants
  <60% | 12.1
  60-80% | 31.4
  >80% | 33.0
  Unknown | 23.5

18. Secondary Outcome: Percentage of Participants With Adequate Quality/Quantity of Tumor Sample
Time Frame: Day 1
Population: All participants enrolled in the study were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 264
percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: This was an epidemiological study with no intervention. Therefore no adverse events were recorded.
Arm/Group | Metastatic Melanoma
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.